CLINICAL TRIAL: NCT02317484
Title: Investigation for Clinical Efficacy and Safety of Ipragliflozin 50mg and 100mg on Type II Diabetes
Acronym: HARUKAS
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Osaka Saiseikai Nakatsu Hospital (Other); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TRIEND1413
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ipragliflozin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ipragliflozin (SGLT2 inhibitor)
  Interventions: Drug: Ipragliflozin (SGLT2 inhibitor)

INTERVENTIONS:
Drug: Ipragliflozin (SGLT2 inhibitor)

SUMMARY:
The purpose of this study is to evaluate clinical efficacy and safety of Sodium Glucose Co-transporter 2 (SGLT2) inhibitor, ipragliflozin, at doses of 50mg and 100mg, for Type II Diabetes under usual care. It is also to investigate and analyze the exploratory influential factor of ipragliflozin treatment on clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes Mellitus, Type 2 patients poorly-controlled by diet and exercise therapies or additional treatment with various diabetic drugs
2. Patients with changes within +- 0.5% of HbA1c
3. Patients with the variation of 6.5% =< HbA1C =<10%
4. Patients with written informed consents
5. Patients whose BMI is =>20kg/m2

Exclusion Criteria:

1. Patients with Diabetes Mellitus, Type 1, other types of diabetes or pregnancy diabetes
2. Patients with history of severe ketoacidosis, diabetic coma or profound coma for the last 6 months
3. Patients with severe infection, in the perioperative period or severe trauma
4. Patients with moderate renal insufficiency (serum creatinine level: male with greater than or equal to 1.5mg/dL、female with greater than or equal to1.3mg/dL)
5. Patients with severe hepatic impairment (judged by the attending doctor)
6. Patients with history of requirement of hospitalization for severe cardiovascular event for the last 6 months of consent
7. Patients in pregnancy, breast-feeding, with childbearing potential or plan of pregnancy
8. Patients with neuropathic bladder or dysuria
9. Patients under treatment with diuretic
10. Patients under SGLT2 treatment at the kickoff point of the study
11. Patients with a history of hypersensitivity to SGLT2 inhibitors
12. Patients who are judged ineligible by the principal investigator

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic and hospital
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11-21 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
HbA1c change level | After 52 weeks from the time of treatment initiation

SECONDARY OUTCOMES:
Sugar metabolism and body composition change levels | After 12, 24, 36, 52 weeks from the time of the start of treatment
  Change levels of the followings after 12, 24, 36, 52 weeks from the time of treatment initiation:
  HbA1c, blood glucose (both at fasting and after eating), glycoalbumin, body weight, BMI, serum lipid (TC、LDL-C、HDL-C、TG), blood pressure (both systolic and diastolic)
HbA1c achievement rate | After 12, 24, 36, 52 weeks from the time of treatment initiation
  The rate of less than HbA1c7.0% achievement after 12, 24, 36, 52 weeks from the time of treatment initiation
Body composition and visceral fat change levels | After 24 and 52 weeks from the time of treatment initiation
  Changes of the body composition examined by DEXA (Dual-energy X-ray absorptiometry) method and visceral fat examined by CT scan after 24 and 52 weeks from the time of treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Haruo Nishimura, Principal Investigator — Osaka Saiseikai Nakatsu Hospital
Locations (1):
- Osaka Saiseikai Nakatsu Hospital, Osaka, Japan